CLINICAL TRIAL: NCT06163755
Title: Comparison of Efficacy of Intra-articular Morphine vs Methylprednisolone in Patients With Knee Osteoarthritis. A Single - Blind, Randomized-controlled Study
Brief Title: Comparison of Efficacy of Intra-articular Morphine vs Methylprednisolone in Patients With Knee Osteoarthritis.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11549
Record Dates: First submitted 2017-12-04; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Methylprednisolone; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group- 1, Morphine Group (Experimental): Morphine 3mg group+0.5% Bupivacaine (total volume 5ml) for Intra-articular knee injection.
  Interventions: Drug: Methylprednisolone 40 MG Injection
- Group- 2 , DepoMedrol ( Methylprednisone) Group (Active Comparator): (control Group - Standard of care ) - DepoMedrol 40mg + 0.25% Bupivacaine (total Volume 5 ml) for Intra-articular knee injection.
  Interventions: Drug: Methylprednisolone 40 MG Injection

INTERVENTIONS:
Drug: Methylprednisolone 40 MG Injection — Intra-articular knee injection will be performed in patient with knee osteoarthritis who meets inclusion criteria. After Random assignment Patient will either get Intra-articular Morphine with Bupivacaine or Depomedrol with Bupivacaine.
  Other Names: Methylprednisolone

SUMMARY:
Prospective randomized double-blind controlled study. Participating patients with knee pain secondary to knee osteoarthritis will be randomized to either the DepoMedrol 40mg + 0.25% Bupivacaine (total Volume 5 ml) vs Morphine 3mg group+0.5% Bupivacaine (total volume 5ml) for their intra-articular knee injection. Before the injections, baseline values of NRS (Numerical rating scale) and WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) Questionnaire will be recorded by investigator. After the injections NRS and WOMAC will be recorded at 30mins and on discharge. Patient will be contacted by phone to assess the effectivity of block or any side effects on day 1, 7,30 and 45, information including NRS (at rest and household activity), WOMAC, supplemental analgesic, Side effects (pruritus, paresthesia, urinary retention, nausea, vomiting, dizziness, rash) will be obtained from the patient at the above time intervals. follow up visit will be scheduled 60days after the procedure for re-evaluation.

DETAILED DESCRIPTION:
It is a randomized prospective single blinded study to be conducted in chronic knee osteoarthritic patients coming to pain clinic with knee pain. Patients will be enrolled in the study after they have been diagnosed with knee pain related to osteoarthritis and conservative management has failed and patient who will meet inclusion criteria, which will include an age ≥ 18 years, patients undergoing intra-articular knee injection for unilateral or bilateral chronic knee pain due to knee osteoarthritis with symptoms (pain, functional limitation due to knee pain and restricted knee range of motion) for a period of at least 3 months in patient who already tried conservative management (Physical therapy and medication management including NSAIDS if there is no contraindication). There is no increased risk to the patients participating in the study therefore the investigators will follow the protocol in the pain clinic for intrarticular knee injections. The investigators will exclude patients with active local or systemic infection (Active Local as well as systemic infection is contraindication for study as there is increase risk of infection into joint space after needling, allergy to any of the medications being used, pregnancy, minors, joint replacement of affected side, coagulopathy (Coagulopathy with INR >1.4, Platelet <100,000, patient with bleeding diathesis, patient on any kind Anti-platelets or anticoagulation medication will be excluded from study as there will be increased risk of bleeding into joint space after needling.), patient refusal, uncontrolled diabetes, blood sugar on day of injection >300mg/dL ( due to increase risk of infection ). Furthermore the patient's vitals will be checked prior to the procedure and standard American Society of Anesthesiology monitors throughout the procedure and for 30 minutes after the procedure. Throughout the study if patient reports uncontrollable pain or any opioid related side effects (which is unlikely with this small dose of medications) then the patient will be asked to follow up with pain clinic. If the patient reports symptomatic hypertension or hyperglycemia related to steroid, they will beasked to return to clinic or to PCP for management. Based on available studies it is unlikely that single, low dose intra-articular morphine injection would cause serious side effects.

The risks, benefits and possible adverse effects will be explained to them and an informed consent obtained. The patients will receive standard care during their pain clinic visit. This includes vital sign assessment, review of current medications, allergies and update of medical history - routinely done on all patients in our clinic. The patient's will be randomized to either the DepoMedrol 40mg vs Morphine 3mg group. Assignment to an arm will be made by selecting from premade envelopes containing random assignments. The patients would undergo an intra-articular knee injection with either steroid or morphine using sterile technique with fluoroscopic guidance which is routine for our practice. Prior to the injection, baseline values of Numerical rating Scale (NRS) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Questionnaire will be recorded by investigator. After the injections NRS and WOMAC will be recorded upon discharge. Patient will be contacted by phone to assess the effectivity of block or any side effects on day 1, 7,30 and 45, telephone call will last for 5-10 minutes, information including NRS (at rest and household activity), WOMAC supplemental analgesic, side effects (pruritus, paresthesia, urinary retention, nausea, vomiting, dizziness, rash) will be obtained from the patient at the above time intervals. Follow up visit will be scheduled 60days after the procedure for re-evaluation and sooner if needed by patient.

Our aim is to assess if the use of morphine will lead to significant pain relief and will lead to promising alternative to currently available steroid medication which have significant serious side effects.

This is a prospective randomized single-blind controlled study. During a 12 months span the investigators treat approximately 24 patients that have knee osteoarthritis and chronic knee pain with an intra-articular knee injection.

The investigators base our sample size on powering the examination of the NRS and WOMAC scores. The investigators estimate the standard deviation of the NRS score at 1.6 and the WOMAC score of 19. If the investigators sample 12 subjects in each of the two injection groups then the test will have 80% power, with a two-sided 0.025 alpha level (two primary outcomes), to detect a difference between NRS scores of 2.08 and WOMAC scores of 24.7. The investigators feel this is a clinically important effect and our sample size is adequate. Additional Information: a. The primary outcome for this study is pain relief, NRS and WOMAC score measured across time on each patient. Also of major importance is the NRS score and WOMAC change from baseline (30 minutes before the procedure) to the final follow-up time point and the follow-up time point containing the lowest score. Furthermore, since this is a randomized study, the investigators assume the baseline WOMAC and NRS should be reasonably similar between the 2 study groups. No prior assumption of non-inferiority has been made. Standard testing is being proposed involving the null hypothesis that the groups are equal.

End Point: #1 Primary end point is the change from the baseline NRS and WOMAC score after 30mins after injection #2 Secondary end point is change from baseline NRS and WOMAC score at 60days (at clinic visit).

Data Analysis:

The maximum pain NRS score and WOMAC decrease from baseline, the pain NRS score and WOMAC score change from baseline to last follow-up. Analgesic consumption over a period of observation will be compared. The two injection groups, steroid vs.morphine, will be compared using Student's t-test, for continuous variables and chi-squared tests for nominal variables. The assumptions of these tests will be examined and data transformations and or nonparametric methods used as indicated. For testing the two primary outcomes (NRS and WOMAC scores) a p-value less than 0.025 will be considered evidence of significance. For the secondary efficacy and safety outcomes, the testing level will be 0.05. The number of patient's in the study would be 24. It is possible that only one of the primary outcomes will show significant differences between the two treatment groups because they are measuring two different domains, pain and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years, patients undergoing intra-articular knee injection for unilateral or bilateral chronic knee pain due to knee osteoarthritis with symptoms (pain, functional limitation due to knee pain and restricted knee range of motion) for a period of at least 3 months in patient who already tried conservative management ( Physical therapy and medication management including NSAIDS if there is no contraindication).

Exclusion Criteria:

We will exclude patients with severe cardiopulmonary or brain disease; active infection; a history of anaphylactic reaction to contrast medium, anesthetic, opioids or steroids; pregnancy; malignant disease, patients who had under gone knee or hip surgery and patients who had been using opioids during the 24 hours prior to the study, patient refusal, uncontrolled diabetes with complications- BS > 300 and patient with ongoing anticoagulation therapy. Patient with osteoarthritis involving joints other than knee causing pain and functional limitation will also be excluded from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC score | 30mins after procedure
  Primary end point is the change from the baseline NRS score after 30mins after injection

SECONDARY OUTCOMES:
NRS score | 30mins after procedure
  Secondary end point is the change from the baseline NRS score after 30mins after injection

IPD SHARING:
Plan to Share IPD: No